CLINICAL TRIAL: NCT06825962
Title: The Effect of Hydration on Postprandial Metabolic Responses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: National Institute for Health Research Leicester Biomedical Research Centre (Unknown)
Responsible Party: Principal Investigator, Lewis James, Dr, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-20370
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Glycaemia
Keywords: Hydration; Dehydration; Hypohydration; Glycemia; Glycaemia; Glucose control
MeSH Terms: conditions — Dehydration | interventions — Drinking

STUDY DESIGN:
Intervention Model Description: Randomised, crossover design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euhydrated (Experimental): Light exercise in a hot environment with water ingested to fully replace sweat losses and maintain euhydration.
  Interventions: Other: Water intake
- Hypohydrated (Experimental): Light exercise in a hot environment with water restricted to induce hypohydration of ~3% body mass through sweating.
  Interventions: Other: Water restriction

INTERVENTIONS:
Other: Water intake — Water ingested to fully replace sweat losses during exercise.
  Arms: Euhydrated
Other: Water restriction — Water restriction to induce hypohydration of ~3% body mass through sweat losses during exercise.
  Arms: Hypohydrated

SUMMARY:
Certain populations, such as industrial workers and endurance athletes are particularly susceptible to dehydration due to exposure to heat for long periods of time causing evaporative water loss via sweating. The physical and cognitive decrements associated with dehydration have been widely researched, however the effect of dehydration on metabolism is lesser known. As climate change is causing temperatures to rise, and metabolic diseases such as type 2 diabetes are more common, the effect of dehydration on metabolism, specifically glycemic response to meals, needs to be established for future recommendations in clinical, environmental and athletic settings.

Therefore, the aim of this study is to investigate the effect of acute exercise-induced dehydration on subsequent metabolic responses to feeding (i.e. glycaemia and insulinaemia).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Generally fit and healthy
* Participate in endurance or intermittent exercise at least 3 times a week or minimum of 150 minutes moderate intensity activity per week

Exclusion Criteria:

* < 18 or > 45
* Any health condition that may affect study outcomes (e.g., endocrine/liver/renal/cardiovascular disease)
* Any morbidity that affects ability to cycle
* Smoker or vaper

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | 6 hours
  Measured using colorimetric assay from venous blood samples

SECONDARY OUTCOMES:
Plasma insulin | 6 hours
  Measured using ELISA from venous blood samples
Plasma osmolality | 6 hours
  Measured using freezing point depression from venous blood samples
Plasma volume change | 6 hours
  Determined from haemoglobin and haematocrit measures in blood samples collected before and after drink ingestion
Urine volume | 6 hours
  Determined from urine samples collected before and after exercise
Body mass | 6 hours
  Determined from weighing participants before and after exercise
Urine specific gravity/osmolality | 6 hours
  Determined from urine samples collected before and after exercise
Thirst sensation | 6 hours
  Measured via 100 mm visual analogue scales 0 mm = not at all thirsty 100 mm = extremely thirsty
Hunger sensation | 6 hours
  Measured via 100 mm visual analogue scales 0 mm = not at all hungry 100 mm = extremely hungry
Fullness sensation | 6 hours
  Measured via 100 mm visual analogue scales 0 mm = not at all full 100 mm = extremely full
Core body temperature | 6 hours
  Measured via ingestible pill
Blood pressure | 6 hours
  Measured via and automated sphygmomanometer

OTHER OUTCOMES:
N-back task for working memory (cognitive function) | 3 hours
  The task will comprise three progressively harder memory loads (1-Back, 2-Back, 3-Back). Each stimulus type will be used in all memory loads. Participants will have to respond using the space bar when they see a stimulus that is presented one, two, or three steps previously, dependent on the load condition. Each phase will comprise 50 trials with ten targets presented centrally on a plain white screen. Each stimulus will be presented for 1000 ms unless the participant responds and in which case the next trial will begin. Commission errors and correct responses will be used as indices of performance. Commission errors occur when participants respond to non-targets.
Go/no-go task for response inhibition (cognitive function) | 3 hours
  Participants will be instructed to press the space bar when an image of a tree appears onscreen ("go" stimulus) and to inhibit responding when an image of a football is presented (the "no-go" stimulus). The task will comprise 200 trials, of which 10% will be no-go trials. Each trial will last 500 ms and will have a black image on a white background. The sequence of stimuli will be the same for each participant. In order to allow for pre-potent tendencies to develop, 50 go trials will precede the first no-go trial. Increased commission error responses (i.e. responding incorrectly on a no-go trial) will indicate reduced response inhibition. Commission errors and correct responses will be measured as indices of performance.
Oculomotor function antisaccade task | 3 hours
  Each trial will start with a 1-second instruction screen prompting participants to focus on the target. A central fixation point will be displayed for one second, followed by a brief blank interval and then the appearance of a red distractor. The distractor will appear randomly to the left or right of the fixation point and will remain visible for 2 seconds. Participants will be instructed to maintain fixation at the centre and then make a saccade in the opposite direction as soon as the distractor appears. The task will include 24 trials, with four additional practice trials. The primary variables measured will be reaction time mean and standard deviation, which reflect inhibition latency and variability. Antisaccade errors, or the number of incorrect saccades, will also be calculated.
Oculomotor function prosaccade task | 3 hours
  Each trial will begin with a 1-second instruction screen, followed by a central fixation point and a brief blank interval. A green target then will appear randomly to the left or right of the fixation point for 2 seconds. Participants will be instructed to fixate at the centre and then make a saccade towards the target. The task will include a total of 14 trials, with four additional practice trials. The variables measured will be reaction time mean and standard deviation, which indicate prosaccade latency and variability.
Oculomotor function smooth pursuit task | 3 hours
  A smooth pursuit task consists of participants following a stimulus with their eyes as it moves in an elliptical pattern on a screen. The stimulus is in motion for 60 seconds. The primary variable measured will be the variability in x and y coordinates of the left and the right eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No